CLINICAL TRIAL: NCT07286825
Title: The Effects of Aromatherapy on Upper Limb Spasticity and Psychosocial Well-being on Stroke Survivors in Residential Care Homes for the Elderly: A Pilot RCT
Brief Title: Aromatherapy on Upper Limb Spasticity on Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Veronica LAI Sze Ki, Assistant Professor, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RD/2024/2.20
Record Dates: First submitted 2025-11-21; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Aromatherapy; Spasticity as Sequela of Stroke
Keywords: aromatherapy massage; stroke survivors; upper limb spasticity
MeSH Terms: interventions — Massage

STUDY DESIGN:
Intervention Model Description: 10-minute massage was given on subjects' upper limbs two times per week by an IFPA aromatherapist using massage oil with a mixture of sweet marjoram essential oil and fractionated coconut organic carrier oil (intervention group) or plain fractionated coconut organic carrier oil (control group) for four weeks.
Who Masked: Participant
Masking Description: Participants are masked for the ingredient of massage oil.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): using massage oil with a mixture of sweet marjoram essential oil and fractionated coconut organic carrier oil
  Interventions: Combination Product: massage oil with a mixture of sweet marjoram essential oil and fractionated coconut organic carrier oil
- Control group (Active Comparator): using massage oil with plain fractionated coconut organic carrier oil
  Interventions: Combination Product: plain fractionated coconut organic carrier oil

INTERVENTIONS:
Combination Product: massage oil with a mixture of sweet marjoram essential oil and fractionated coconut organic carrier oil — 10-minute massage was given on subjects' upper limbs two times per week by an IFPA aromatherapist using massage oil with a mixture of sweet marjoram essential oil and fractionated coconut organic carrier oil.
  Arms: Intervention group
Combination Product: plain fractionated coconut organic carrier oil — 10-minute massage was given on subjects' upper limbs two times per week by an IFPA aromatherapist using plain fractionated coconut organic carrier oil as massage oil.
  Arms: Control group

SUMMARY:
This study employed a double-arm, pre- and post-test design. Stroke survivors aged 65 or above with post-stroke upper limbs spasticity were recruited from two RCHEs in Hong Kong between February and June 2025, and were divided into control and intervention groups. 10-minute massage was given on subjects' upper limbs two times per week by an IFPA aromatherapist using massage oil with a mixture of sweet marjoram essential oil and fractionated coconut organic carrier oil (intervention group) or plain fractionated coconut organic carrier oil (control group) for four weeks. The range of motion (ROM) of the upper limbs in three planes, i.e., abduction, flexion and extension and pain level and blood pressure were assessed before and after each massage session. Psychosocial well-being of elders was assessed at baseline and 4 weeks post-intervention using Generalised Anxiety Disorder (GAD-7) and Patient Health Questionnaire (PHQ-9).

DETAILED DESCRIPTION:
Study design This study employed a double-arm, pre- and post-test design. The study was conducted in two RCHEs in Hong Kong under a non-government organisation, Po Leung Kuk (PLK).

Participants We took reference from a pilot RCT on the effect of aromatherapy acupressure on hemiplegic shoulder and motor power among stroke patients recruited 30 patients (15 control and 15 intervention) (Shin & Lee, 2007). In our study, 30 elders aged 65 or above with post-stroke upper limbs spasticity were recruited from two RCHEs in Hong Kong and evenly divided in both control and intervention groups (please refer to CONSORT flowchart in Fig. 2). Among both groups, only two elders from the control group dropped out due to admission to hospital during the research period. Participants were considered eligible if: (1) he/she is communicable with either Chinese or English, and (2) suffering from upper-limb post-stroke spasticity. In addition, participants will be excluded if: (1) he/she is currently receiving aromatherapy massage therapies, (2) he/she has external wound on the massage areas.

An information sheet was given, and consent was sought from each carer and elder before the intervention. All elders and carers were free to withdraw consent at any time. Where possible, clarification on the specific area of withdrawal, but not obligatory. Previously collected data was use in the analyses.

Procedures A 10-minute massage was given on elders' upper limbs two times per week by an IFPA aromatherapist using massage oil with a mixture of sweet marjoram essential oil and fractionated coconut organic carrier oil (intervention group) or plain fractionated coconut organic carrier oil (control group) for four weeks (8 sessions in total). Massage steps and rhythm and intensity are standardised for all subjects. Range of motion (ROM) and pain level was measured before and after each session of massage and psychosocial well-being will be measured at baseline and 4 weeks after the intervention.

Upper limb massage steps were standardized as follow:

Effleurage was done on the upper limbs and shoulders with mild pressure using hands, which mould themselves to the shape of the body being massaged (Price et al., 2020). 5-Step massage was done with sweet marjoram massage oil on both upper limbs as well as shoulders (as shown below). Whole massage process lasted for 10-15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* he/she is communicable with either Chinese or English, and
* suffering from upper-limb post-stroke spasticity

Exclusion Criteria:

* he/she is currently receiving aromatherapy massage therapies
* he/she has external wound on the massage areas.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Range of motion (ROM) on shoulder joints | Before and after each massage session for 4 weeks in total
  Range of motion (ROM) will be assessed on shoulder joints as the primary outcome. The shoulder complex consists of four joints: the glenohumeral (GH), sternoclavicular (SC), acromioclavicular (AC) and scapulothoracic joints. The ROM of shoulder requires coordinated motion of all these joint. To evaluate the functional ROM of the shoulder, a goniometer will be used for measuring the passive or active ROM values (degrees) before and after each week of massage for 4 weeks in total. Abduction, flexion and extension ROM will be measured.

SECONDARY OUTCOMES:
The Chinese Version of Generalised Anxiety Disorder (GAD-7) | Week 0 and Week 4 after completing all massage sessions
  The Chinese version of GAD-7 will be used for assessing the anxiety level severity in clinical practice (Spitzer et al., 2006). It consists of seven items; each item is scored from 0 to 3 with the total score ranges from 0 to 21. The internal consistency of the GAD-7 was excellent (Cronbach' α = .92).
Patient Health Questionnaire (PHQ-9) | Week 0 and Week 4 after completing all massage sessions
  The Chinese version of PHQ-9, which is widely used in different community settings for depression screening, will be used. PHQ-9 consists of nine-item depression module with internal consistency (Cronbach' α) of α =0.87.

CONTACTS AND LOCATIONS:
Overall Officials: Sze Ki Veronica LAI, Dr, Principal Investigator — School of Nursing and Health Studies, Hong Kong Metropolitan Universit
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The researchers will guarantee full confidentiality. All data will be kept 2 years after the project completion date. All soft copies of data will be destroyed by reformatting the disk (destroying everything on it). Hard copies will be destroyed by shredding then cross shredding.